CLINICAL TRIAL: NCT03500419
Title: Penile Length Maintenance Post-Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew (Matt) J. Ziegelmann, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-001013
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer; Penile Diseases
MeSH Terms: conditions — Prostatic Neoplasms; Penile Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Active Comparator): No treatment will be administered for the initial 6 months post-prostatectomy. This is necessary as a measure to review post-prostatectomy penile length changes.
  Interventions: Other: No treatment
- Group AB - PTT 1-2x daily x 5-7 days/week x 5 months (Experimental): Men will utilize penile traction therapy for 30 minutes 1-2 times daily, 5-7 times a week, beginning 4 weeks post-prostatectomy. Men will remain in this phase for a period of 5 months.
  Interventions: Device: RestoreX

INTERVENTIONS:
Device: RestoreX — PTT - Penile traction therapy in the straight position.
  Arms: Group AB - PTT 1-2x daily x 5-7 days/week x 5 months
Other: No treatment — Control group. No treatment will be given for the 6 months post-prostatectomy
  Arms: Control

SUMMARY:
The objective of the current study is to evaluate the efficacy of a novel, class I (ie. lowest risk, clinical studies not required) medical penile traction device in preventing loss of penile length in men undergoing robotic-assisted prostatectomy.

DETAILED DESCRIPTION:
The treatment of prostate cancer results in several known sexual dysfunctions, including erectile dysfunction, orgasmic dysfunction, ejaculatory dysfunction, penile curvature (Peyronie's disease), and reduced penile length. Among the dysfunctions, loss of penile length is often one that results in significant distress and bother to patients. Beyond the esthetic concerns, reduced penile length may lead to inability to participate in sexual intercourse, difficulty with future interventions to restore erectile function, and lead to worsened urinary hygiene.

Penile traction therapy (PTT) is currently the best available treatment to maintain or restore lost penile length due to conditions that reduce length. To date, no studies have evaluated the benefits of using PTT in this clinical setting. The objective of the current study is to evaluate the efficacy of a novel penile traction device (RestoreX®), created and funded through Mayo Ventures, in maintaining or restoring reduced penile length.

To accomplish the study, a population of men from Mayo Clinic who have undergone a prostatectomy will be enrolled and randomized to utilize the device for varying amounts of time. Outcomes will be assessed at 6 and 9 months post-prostatectomy and results are to be used with the intent to publish in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing robotic prostatectomy
* Seen in the post-prostatectomy rehab clinic

Exclusion Criteria:

• Urethral complications from prostatectomy at the time of baseline visit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ziegelmann, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No treatment was administered for the initial 6 months post-prostatectomy. This is necessary as a measure to review post-prostatectomy penile length changes.
  No treatment: Control group. No treatment was given for the 6 months post-prostatectomy
- PTT 1-2x Daily x 5-7 Days/Week x 5 Months: Men utilized penile traction therapy for 30 minutes 1-2 times daily, 5-7 times a week, beginning 4 weeks post-prostatectomy for a period of 5 months.
  RestoreX: PTT - Penile traction therapy in the straight position.
Period: Overall Study
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Started | 27 | 55
Completed | 25 | 30
Not Completed | 2 | 25
Not completed — Withdrawal by Subject | 2 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months | Total
Number analyzed (Participants) | 27 | 55 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (4.5) | 58.7 (6.8) | 58.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 55 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 25 | 48 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 27 | 55 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change in Penile Length
Description: Stretched penile length measured in centimeters from pubic symphysis to glanular corona
Time Frame: Baseline, 6 months
Population: 6 months data was not collected nor analyzed for 2 subjects in control arm and 25 subjects in PTT arm.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Number analyzed (Participants) | 25 | 30
centimeters | 0.3 (1.5) | 1.6 (1.0)

2. Secondary Outcome: Erectogenic Therapy Use
Description: The percentage of subjects to use a phosphodiesterase-5 inhibitor for erectogenic therapy use
Time Frame: 6 months
Population: 6 months data was not collected nor analyzed for 2 subjects in control arm and 25 subjects in PTT arm.
Measure: Number; unit: percentage of subjects
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Number analyzed (Participants) | 25 | 30
percentage of subjects | 94 | 86

3. Secondary Outcome: Intracavernosal Injections
Description: The percentage of subjects to use intracavernosal injections
Time Frame: 6 months
Population: 6 months data was not collected nor analyzed for 2 subjects in control arm and 25 subjects in PTT arm.
Measure: Number; unit: percentage of subjects
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Number analyzed (Participants) | 25 | 30
percentage of subjects | 50 | 19

4. Secondary Outcome: Change in Erectile Function Domain of International Index of Erectile Function (IIEF)
Description: Erectile function domain will be measured by using the International Index of Erectile Function (IIEF) questionnaire. IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
Time Frame: baseline, 6 months
Population: 6 months data was not collected nor analyzed for 2 subjects in control arm and 25 subjects in PTT arm. Negative denotes loss of function.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Number analyzed (Participants) | 25 | 30
units on a scale | -6.5 [-21.5 to -2] | 0 [-7.5 to 4]

5. Secondary Outcome: Change in Intercourse Satisfaction Domain of International Index of Erectile Function (IIEF)
Description: Intercourse satisfaction will be measured by using the International Index of Erectile Function (IIEF) questionnaire. IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
Time Frame: Baseline, 6 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Number analyzed (Participants) | 25 | 30
units on a scale | -3.5 [-7.0 to 0] | 1 [-2 to 7]

6. Secondary Outcome: Change in Overall Satisfaction Domain of International Index of Erectile Function (IIEF)
Description: Overall satisfaction domain will be measured by using the International Index of Erectile Function (IIEF) questionnaire. IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
Time Frame: Baseline, 6 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
Number analyzed (Participants) | 25 | 30
units on a scale | -3 [-6 to -1] | 0 [-2.8 to 0.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until end of intervention, approximately 6 months.
Arm/Group | Control | PTT 1-2x Daily x 5-7 Days/Week x 5 Months
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/55
Other Adverse Events (participants affected / at risk) | 0/27 | 17/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=27) | PTT 1-2x Daily x 5-7 Days/Week x 5 Months (N=55)
Temporary penile erythema or discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Temporary mile penile discomfort (General disorders) | 0 (0) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03500419/Prot_SAP_002.pdf